CLINICAL TRIAL: NCT01425619
Title: The Effect of Medical Clowns and Topical Anesthetic Cream on Pain and Anxiety in Children Undergoing Allergy Skin Tests
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Meir Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: CLOWN 1
Record Dates: First submitted 2011-08-21; First posted 2011-08-30 (Estimated); Last update posted 2015-10-08 (Estimated); Status verified 2012-09

CONDITIONS: Anxiety Disorder; Allergic Skin Reaction
Keywords: Anxiety Disorder due to Allergy Skin Testing
MeSH Terms: conditions — Anxiety Disorders | interventions — Cetomacrogol

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Placebo cream, Skin test, Anxiety, Pain (Placebo Comparator): After placing a placebo cream on both arms, pain and anxiety resulting from performing allergy skin test on one of the arms will be evaluated
  Interventions: Biological: Cream of Macrogol cetostearyl ethers
- Anesthetic cream, pain and anxiety, skin test (Active Comparator): After placing a placebo cream on one arm and anesthetic cream on the second arm, pain and anxiety resulting from performing allergy skin test on the second arm will be evaluated
  Interventions: Drug: Cream of Lidocaine 2.5 %.and Prilocaine 2.5 %
- Medical clown, placebo cream, skin test (Active Comparator): After placing a placebo cream on both arms and after receiving care and treatment from a medical clown, pain and anxiety resulting from performing allergy skin test on one of the arms will be evaluated
  Interventions: Behavioral: Care and treatment from a medical clown
- Medical clown, Anesthetic cream, Skin test (Active Comparator): After placing a placebo cream on one arm and anesthetic cream on the second arm and after receiving care and treatment from a medical clown, pain and anxiety resulting from performing allergy skin test on the second arm will be evaluated
  Interventions: Behavioral: Care and treatment from a medical clown

INTERVENTIONS:
Biological: Cream of Macrogol cetostearyl ethers — The cream will be applied on the volar aspect of both arms for 1 hour
  Other Names: Cetomacrogol
  Arms: Placebo cream, Skin test, Anxiety, Pain
Drug: Cream of Lidocaine 2.5 %.and Prilocaine 2.5 % — 1-2 gr. of the cream will be applied on the volar aspect of the second arm; for 1 hour
  Other Names: EMLA 5%
  Arms: Anesthetic cream, pain and anxiety, skin test
Behavioral: Care and treatment from a medical clown — Medical clown will entertain the children before, during and after performing the skin test. Placebo cream will be applied on both arms.
  Arms: Medical clown, placebo cream, skin test
Behavioral: Care and treatment from a medical clown — Medical clown will entertain the children, placebo cream will be applied on one arm and anesthetic cream on the second arm
  Arms: Medical clown, Anesthetic cream, Skin test

SUMMARY:
Allergy skin tests are occasionally associated with pain and anxiety in patients undergoing this procedure. The investigators intend to examine if medical clowns compared with local anesthetic cream can decrease these feelings in children.

ELIGIBILITY:
Inclusion Criteria:

* Any child undergoing allergy prick skin test

Exclusion Criteria:

* Children suffering from coulrophobia (phobia of clowns)
* Children with a known hypersensitivity to EMLA 5% cream
* Children who have undergone a painful medical procedure (surgery, dental procedures, blood drawing) over the past 3 months
* Children who, for medical reasons, must have their skin test performed on an area other than the volar aspect of the arm

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 160 (Estimated)
Dates: Start 2011-10; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
The level of anxiety experienced by children undergoing allergy skin tests and receiving application of local anesthetic cream and/or care and treatment from medical clowns | 1.5 hour

SECONDARY OUTCOMES:
Severity of pain experienced by these children | 1.5 hour

CONTACTS AND LOCATIONS:
Locations (1):
- Arnon Goldberg, Allergy and Clinical Immunology Unit, Meir Medical Center, Kfar Saba, Israel